CLINICAL TRIAL: NCT04047537
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Metabolic Effects of Two Formulations of a Food Product (WBF-0011) When Administered to Subjects With Type 2 Diabetes Treated With Diet and Exercise Alone or in Combination With Metformin
Brief Title: Placebo-Controlled Clinical Nutrition Study of the Metabolic Effects of Food Product WBF-0011 in Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid interference
Sponsor: Pendulum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AFCRO-104
Record Dates: First submitted 2019-07-26; First posted 2019-08-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: WBF-0011 (Other): 2 capsules/day (one in the morning and one in the evening), taken with meal for 12 weeks
  Interventions: Other: Medical Food Formulation 1
- Experimental: WBF-0011 (0.2X concentration) (Other): 2 capsules/day (one in the morning and one in the evening), taken with meal for 12 weeks
  Interventions: Other: Medical Food Formulation 2
- Placebo (Other): 2 capsules/day (one in the morning and one in the evening), taken with meal for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Medical Food Formulation 1 — WBF-0011
  Arms: Experimental: WBF-0011
Other: Medical Food Formulation 2 — WBF-0011 (0.2X concentration)
  Arms: Experimental: WBF-0011 (0.2X concentration)
Other: Placebo — Placebo Capsules identical to those containing Formulation 1 and 2
  Arms: Placebo

SUMMARY:
This 12 week placebo-controlled study evaluates the safety and impact of 2 different strengths of the medical food formulation WBF-0011.

DETAILED DESCRIPTION:
The medical food formulations being tested in this study contain butyrate-producing organisms plus a microbial strain that contributes to the integrity of the colonic mucin barrier. The microbes have been fully characterized, certified as Generally Recognized As Safe (GRAS) and manufactured to Good Manufacturing Practice (GMP) standards using excipients that are also GRAS qualified.

Subjects will receive their randomized formulation twice a day for 12 weeks.The target population will be patients with Type 2 Diabetes who are not treated with anti-diabetic agents or are treated with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent
* Have type 2 diabetes treated with diet and exercise alone or in combination with metformin
* If treated with metformin, must have been on a stable dose of the drug for a minimum of 3 months with a stable A1c value
* If treated with diet and exercise alone, must have A1c value ≥6.5%
* If treated with diet and exercise + metformin, must have a stable A1c between 7.0% and 8.5% for at least 3 months
* BMI >25 but <45
* If female, must meet all the following criteria:

  1. Not pregnant or breastfeeding
  2. If of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice and be willing to continue to practice appropriate birth control during the entire duration of the study
* Must be able to communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

* Subjects who have received an antibiotic, antifungal, antiparasitic, or antiviral treatment within 30 days prior to study entry
* Subjects who plan to use antibiotic, antifungal, antiparasitic, or antiviral treatment during the study
* Subjects using a proton pump inhibitor must be on a consistent dose that will be maintained throughout the study period
* Present use of probiotics/nutritional supplements. (Note: The use of replacement doses of Vitamin D, calcium supplements, and a single daily multi-vitamin tablet is allowed)
* Subjects who have participated in a structured weight-loss program within the past 3 months
* Subjects who have changed body weight ≥3% within the past month
* Excess alcohol consumption; with an alcoholic drink defined as 284 ml of beer, lager, stout , 100 ml of wine or 35.5 ml spirits

  1. Women: More than 11 standard drinks/week
  2. Men: More than 17 standard drinks/week
* Subjects who have received an experimental drug within 30 days prior to study entry
* Hospitalization for any reason within the 3 months prior to study entry (Same day surgery centre visits/procedures allowed)
* Active GI disease
* History of any surgery on the gastrointestinal tract except appendectomy and cholecystectomy
* Cystic fibrosis
* Significant renal Impairment defined as estimated Glomerular Filtration Rate <45 ml/min
* Subjects receiving systemic corticosteroid therapy
* Subjects receiving Immunosuppression therapy
* Subjects with any condition that the investigator deems as a sound reason for disqualification from enrollment into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | From Baseline to Week 12
  Change from baseline to Week 12 in each of the treatment groups as compared to placebo in A1c levels

SECONDARY OUTCOMES:
3-hour blood glucose Area Under the Curve (AUC) | Baseline to Weeks 2, 6, 9 and 12
  as measured by the Continuous Glucose Monitor (CGM) device in clinic during standardized 3-hour Meal Tolerance Test (MTT)
3-hour plasma glucose AUC | Baseline to Weeks 2, 6, 9 and 12
  as measured by laboratory plasma glucose measurements during standardized 3-hour Meal Tolerance Test (MTT)
3-hour blood glucose AUC | Baseline to Weeks 1, 3, 4, 5, 7, 8, 10, and 11.
  as measured by the CGM device at home during standardized 3-hour Meal Tolerance Test (MTT)
24-hour CGM | From Baseline to Week 12
  Time in range (70 to 180 mg/dL)/24-hour period
Fasting Lipid Panel | From Baseline to Week 12
  Change in fasting serum concentrations of total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides
Body weight | From Baseline to Week 12
  Change in body weight in kilograms
Adverse Events | From Baseline to Week 12
  Number of participants with adverse events related to therapy
Change from baseline in Laboratory Chemistry Values | From Baseline to Week 12
  Number of Participants With Abnormal Laboratory Values Related to Therapy
Change from baseline in Laboratory Complete Blood count Values | From Baseline to Week 12
  Number of Participants With Abnormal Laboratory Values Related to Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Orville Kolterman, MD, Study Director — Whole Biome
Locations (1):
- Atlantia Food Clinical Trials, 1st Floor, Block C, Heron House, Blackpool Retail Park, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No